CLINICAL TRIAL: NCT05863117
Title: Syphilis and HIV Point of Care Testing (POCT) to Improve Access to Testing Among Inner City, Remote, Rural and Hard to Reach Populations in Saskatchewan
Brief Title: Syphilis and HIV Point of Care Testing (POCT) in Saskatchewan
Acronym: SHIVER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wellness Wheel Medical Clinic (Other)
Collaborators: CIHR Canadian HIV Trials Network (Network); University of Saskatchewan (Other); Saskatchewan Health Authority - Regina Area (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: NFL-CBD-0
Record Dates: First submitted 2023-04-19; First posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Syphilis; HIV Infections
Keywords: point of care testing
MeSH Terms: conditions — Syphilis; HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Reveal Rapid TP (from MedMira) — Point of care tests for HIV and Syphilis
  Other Names: INSTI HIV-1/2 HIV test; INSTI Multiplex HIV-1/2 Syphilis

SUMMARY:
The goal of this clinical trial is to learn about Syphilis and HIV point of care testing among inner city, remote, rural and hard to reach populations in Saskatchewan. The main question[s] it aims to answer are:

1. To evaluate the field diagnostic test performance (e.g. sensitivity, specificity, predictive values) of finger prick whole blood point of care testing (POCT) when compared to standard serum based testing for syphilis POCT, HIV POCT and dual syphilis and HIV POCT.
2. To evaluate the clinical utility of POCT for the prompt management and public health follow up of syphilis and HIV cases as compared to usual testing, specifically:

   1. Time to diagnosis
   2. Time to treatment
   3. Number of contacts exposed to untreated infections
   4. For HIV diagnoses, time to connection to clinical provider for ongoing management of HIV
3. To evaluate the acceptability and feasibility of POCT among different populations for syphilis and HIV among at risk and/or hard to reach populations, specifically:

   1. Health care provider experiences of feasibility and acceptability of the POCT used in this pilot
   2. Client acceptability and experiences with POCT in this pilot
   3. Client preferences for test offered (syphilis only, HIV only, or dual test of HIV and syphilis 4. To evaluate the acceptability and feasibility of syphilis alone, HIV alone or combined syphilis/HIV POCT among at-risk and/or hard to reach populations.

Participants will be assessed for risk factors that may increase risk of infectious disease such as substance use and sexual habits. They will then be offered a choice of 1 of 3 POCT(Syphilis alone, HIV alone or a dual HIV/Syphilis test). Serology will be obtained for sexually transmitted and blood born infections (STBBI's) and then the point of care test (POCT) will be completed. Following the testing the participant will complete a short survey on their experience.

ELIGIBILITY:
Inclusion Criteria:

* 1650 consecutive individuals
* > 16 years accessing STBBI testing at specific locations and able to provide informed consent. PLWH and persons who are syphilis positive may also eligible to participate.

Exclusion Criteria:

° Less than 16 years, unable to provide signed informed consent (e.g., intoxicated)

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1650 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Syphilis-Comparison between point of care testing and serology testing for Syphilis and HIV | 12-18 months
  To evaluate the field diagnostic test performance of finger prick whole blood point of care testing (POCT) when compared to standard serum based testing for syphilis POCT.
HIV- Comparison between point of care testing and serology testing for Syphilis and HIV | 12-18 months
  HIV- To evaluate the field diagnostic test performance of finger prick whole blood point of care testing (POCT) when compared to standard serum based testing for HIV POCT.
Syphilis/HIV- Comparison between point of care testing and serology testing for Syphilis and HIV | 12-18 months
  Dual HIV/Syphilis-To evaluate the field diagnostic test performance of finger prick whole blood point of care testing (POCT) when compared to standard serum based testing for dual syphilis and HIV POCT.

SECONDARY OUTCOMES:
Time to diagnosis-Clinical utility of POCT for management and follow up of Syphilis and HIV | 12-18 months
  To evaluate the clinical utility of POCT for the prompt management and public health follow up of syphilis and HIV cases as compared to usual testing, specifically: Time to diagnosis
Evaluate the acceptability and feasibility of POCT for syphilis and HIV | 12-18 months
  To evaluate the acceptability and feasibility by using a patient experience survey of POCT among different populations for syphilis and HIV among at risk and/or hard to reach populations, specifically: Health care provider experiences of feasibility and acceptability of the POCT used in this pilot b) Client acceptability and experiences with POCT in this pilot c) Client preferences for test offered (syphilis only, HIV only, or dual test of HIV and syphilis
HIV-Comparison of acceptability and feasibility by using a patient experience survey of syphilis alone, HIV alone and dual HIV/Syphilis point of care testing among different populations. | 12-18 months
  To evaluate the acceptability and feasibility of HIV alone among at-risk and/or hard to reach populations
Dual HIV/Syphilis-Comparison of acceptability and feasibility by using a patient experience survey of syphilis alone, HIV alone and dual HIV/Syphilis point of care testing among different populations. | 12-18 months
  To evaluate the acceptability and feasibility of combined syphilis/HIV POCT among at-risk and/or hard to reach populations
Syphilis-Comparison of acceptability and feasibility by using a patient experience survey of syphilis alone, HIV alone and dual HIV/Syphilis point of care testing among different populations. | 12-18 months
  To evaluate the acceptability and feasibility of syphilis alone, among at-risk and/or hard to reach populations
Time to treatment-Clinical utility of POCT for management and follow up of Syphilis and HIV | 12-18 months
  To evaluate the clinical utility of POCT for the prompt management and public health follow up of syphilis and HIV cases as compared to usual testing, specifically:Time to treatment
Number of contacts-Clinical utility of POCT for management and follow up of Syphilis and HIV | 12-18 months
  To evaluate the clinical utility of POCT for the prompt management and public health follow up of syphilis and HIV cases as compared to usual testing, specifically: Number of contacts exposed to untreated infections
Time to connection-Clinical utility of POCT for management and follow up of Syphilis and HIV | 12-18 months
  To evaluate the clinical utility of POCT for the prompt management and public health follow up of syphilis and HIV cases as compared to usual testing, specifically: For HIV diagnoses, time to connection to clinical provider for ongoing management of HIV.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Skinner, MD, Principal Investigator — Saskatchewan Health Region
Locations (2):
- Canada (2):
  - Queen City Wellness Pharmacy, Regina, Saskatchewan
  - Wellness Wheel Medical Clinic, Regina, Saskatchewan

IPD SHARING:
Plan to Share IPD: No